CLINICAL TRIAL: NCT01891071
Title: Lung Volume Recruitment for Lung Function and Cough Impairment in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-LVR-01; 20120570-01H (Other: Ottawa Hospital Research Ethics Board); AA-HCLM-14-019 (Other: Comité d'éthique de la recherche du Centre de santé et services sociaux Champlain-Charles LeMoyne)
Record Dates: First submitted 2013-02-25; First posted 2013-07-02 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Lung volume recruitment; Pulmonary function impairment; Cough impairment
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lung volume recruitment (Experimental): Lung volume recruitment twice daily for 9 months
  Interventions: Procedure: Lung volume recruitment
- Standard care (No Intervention): Standard care

INTERVENTIONS:
Procedure: Lung volume recruitment — Inflation of the lungs to their maximal insufflation capacity by the consecutive delivery, by a manual resuscitator in this study, of volumes of air that are held with a closed glottis
  Other Names: Air stacking; Glossophayngeal breathing
  Arms: Lung volume recruitment

SUMMARY:
Multiple sclerosis is a neurological disease that can affect lung function and cough efficacy. This pilot study will examine whether the lung volume recruitment technique can slow down the decline in lung function and cough.

ELIGIBILITY:
Inclusion Criteria:

* History of multiple sclerosis, diagnosed by a neurologist in accordance with the 2010 McDonald criteria

Exclusion Criteria:

* Concomitant parenchymal pulmonary disease or pleural disease
* Symptomatic cardiomyopathy
* Unable to perform pulmonary function testing or lung volume recruitment, due to comprehension or cooperation issues, physical inability such as bulbar or cerebellar dysfunction
* Contra-indication to pulmonary function testing or lung volume recruitment such as myocardial infarction, bleeding aortic aneurysm, intracranial hemorrhage within the previous month
* Known susceptibility to pneumothorax or pneumomediastinum
* Not competent to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Rate of decline of FVC (forced vital capacity) | up to 9 months

SECONDARY OUTCOMES:
Rate of decline of peak cough flow | baseline, 2, 4, 6 and 9 months
Change from baseline in FVC at 2, 4, 6 and 9 months | baseline vs 2, 4, 6 and 9 months
Change from baseline in peak cough flow at 2, 4, 6 and 9 months | baseline vs 2, 4, 6 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Nadim Srour, MD, MSc, Study Chair — Université de Sherbrooke; Douglas A McKim, MD, Principal Investigator — The Ottawa Hospital
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Hôpital Charles-LeMoyne, Greenfield Park, Quebec

REFERENCES:
- [Background] Srour N, LeBlanc C, King J, McKim DA. Lung volume recruitment in multiple sclerosis. PLoS One. 2013;8(1):e56676. doi: 10.1371/journal.pone.0056676. Epub 2013 Jan 31. PMID 23383293